CLINICAL TRIAL: NCT06353139
Title: Modified Olfactory Training for Patients With Olfactory Disfunction:A Randomized Clinical Trial
Brief Title: The Efficacy of Modified Olfactory Training for Patients With Olfactory Dysfunction
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Principal Investigator, Dawei Wu, Associate Researcher, Peking University Third Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 90591
Record Dates: First submitted 2024-03-30; First posted 2024-04-08 (Actual); Last update posted 2024-04-08 (Actual); Status verified 2024-04

CONDITIONS: Olfactory Impairment
MeSH Terms: conditions — Olfaction Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The traditional olfactory training (Active Comparator)
  Interventions: Device: Modified olfactory training device
- The modified olfactory training (Experimental)
  Interventions: Device: Modified olfactory training device

INTERVENTIONS:
Device: Modified olfactory training device — Conduct olfactory training in patients with olfactory disorders

SUMMARY:
The goal of this clinical trial is to validate the effectiveness of the modified olfactory training device, the main questions it aims to answer are:

Is it possible that the device can treat olfactory disorders in adults? Compared to the conventional device, how efficient is the modified olfactory training device for treating patients with olfactory disfunction?

DETAILED DESCRIPTION:
Olfactory training is a new therapy that improves olfactory function by exposing patients to various types of odors through regular, repetitive active sniffing. However, there are still many problems with olfactory training in clinical practice, including poor patient adherence, lack of standardized and uniform procedures, and inconvenient carrying of devices.

Now, the investigators have initially developed an olfactory training device based on expiratory pressure, and the advantages of the improved device are as follows: bi-directional airflow, positive pressure and the function of voice prompts and automatic counting.

In this study, the investigators planned to recruit 72 patients and divided them into two groups for olfactory training with conventional and modified devices, and validate the effectiveness of the modified device based on the comparison of the outcomes of the two groups.

ELIGIBILITY:
Inclusion Criteria:

1. Patients diagnosed with olfactory disorder when TDI score was less than 30.75.
2. Patients would perform Sniffin' Sticks examination.
3. Voluntarily sign the informed consent form
4. Able to undergo olfactory training and participate in follow-up visits

Exclusion Criteria:

1. Smoking
2. Combined with chronic diseases, such as hypertension, diabetes, bronchopneumonia, chronic obstructive pulmonary disease, etc.
3. Those who have taken oral glucocorticoids, antibiotics, anti-leukotrienes, and antihistamines within four weeks will be excluded.
4. Patients who cannot tolerate olfactory function testing and treatment
5. Severe coexisting diseases: such as malignant tumors, life expectancy <2 years
6. Patients who are pregnant or planning to become pregnant
7. According to the researcher's judgment, the patient is unable to complete this study or cannot comply with the requirements of this study (such as memory or behavioral abnormalities, depression, heavy drinking, past breach of contract)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2023-07-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Clinically significant olfactory improvement | 1 year
  a clinically significant olfactory improvement as measured by Sniffin' Sticks threshold, discrimination, and identification（TDI)( more than 6 scores)

CONTACTS AND LOCATIONS:
Locations (1):
- Dawei Wu, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No
We will decide whether to share the individual participant data after the study.

REFERENCES:
- [Result] Yuan F, Huang T, Wei Y, Wu D. Steroids and Olfactory Training for Postviral Olfactory Dysfunction: A Systematic Review. Front Neurosci. 2021 Aug 12;15:708510. doi: 10.3389/fnins.2021.708510. eCollection 2021. PMID 34456675
- [Result] Patel ZM, Holbrook EH, Turner JH, Adappa ND, Albers MW, Altundag A, Appenzeller S, Costanzo RM, Croy I, Davis GE, Dehgani-Mobaraki P, Doty RL, Duffy VB, Goldstein BJ, Gudis DA, Haehner A, Higgins TS, Hopkins C, Huart C, Hummel T, Jitaroon K, Kern RC, Khanwalkar AR, Kobayashi M, Kondo K, Lane AP, Lechner M, Leopold DA, Levy JM, Marmura MJ, Mclelland L, Miwa T, Moberg PJ, Mueller CA, Nigwekar SU, O'Brien EK, Paunescu TG, Pellegrino R, Philpott C, Pinto JM, Reiter ER, Roalf DR, Rowan NR, Schlosser RJ, Schwob J, Seiden AM, Smith TL, Soler ZM, Sowerby L, Tan BK, Thamboo A, Wrobel B, Yan CH. International consensus statement on allergy and rhinology: Olfaction. Int Forum Allergy Rhinol. 2022 Apr;12(4):327-680. doi: 10.1002/alr.22929. PMID 35373533